CLINICAL TRIAL: NCT04679116
Title: Laparoscopic vs Open Bilateral Inguinal Hernia Repair
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: General Hospital of Larissa (Other)
Responsible Party: Principal Investigator, Georgios Koukoulis, General Surgery Consultant, General Hospital of Larissa
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1726
Record Dates: First submitted 2020-12-11; First posted 2020-12-22 (Actual); Last update posted 2021-02-03 (Actual); Status verified 2021-02

CONDITIONS: Inguinal Hernia Bilateral
Keywords: bilateral inguinal hernia repair

STUDY DESIGN:
Intervention Model Description: prospective, non randomised
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Laparoscopic (Other): laparoscopic inguinal hernia repair, TAPP
  Interventions: Procedure: Laparoscopic bilateral inguinal hernia repair
- Open (Other): open inguinal hernia repair
  Interventions: Procedure: Open bilateral inguinal hernia repair

INTERVENTIONS:
Procedure: Laparoscopic bilateral inguinal hernia repair — Laparoscopic bilateral inguinal hernia repair
  Arms: Laparoscopic
Procedure: Open bilateral inguinal hernia repair — Open bilateral inguinal hernia repair
  Arms: Open

SUMMARY:
The European Hernia Society Guidelines of 2018 suggest that laparoscopic surgery should be preferred over open surgery for bilateral inguinal hernia repair even though scientific evidence are scarce. We will conduct a prospective, non randomise control trial, to investigate the superiority of one technique over the other.

ELIGIBILITY:
Inclusion Criteria:

* bilateral inguinal hernia

Exclusion Criteria:

* American Society of Anaesthesiology score >3
* complicated inguinal hernias

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 100 (Estimated)
Dates: Start 2021-01-02 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Post operative Pain | 24 hours post surgery
  Evaluation of the post operative pain 24 hours after surgery. For the assessment of the pain will be used the Visual Analog Scale (VAS) score. (VAS Score Scale from 0-10, 0 no pain, 10 max pain)

SECONDARY OUTCOMES:
days of hospitalization | 30 days
  days that need to be hospitalised after surgery
urinary retention | 8 hours
  inability to voluntarily void urine up to 8 hours post surgery
complications | 30 days
  presence of surgery related complications
recurrence | 1 year
  recurrence of one or two of the hernias treated at the clinical evaluation one year after surgery
chronic pain | 1 year
  For the evaluation of the chronic pain will be used the registry for abdominal wall hernias Quality of Life questionnaire (EuraHS QoL) scale from 0 to 10. (0 = no pain 10=worst pain imaginable)
foreign body sensation to the inguinal area | 1 year
  For the evaluation of the foreign body sensation to the inguinal area will be used the Carolinas Comfort Scale (scale from 0 to 5, 0= no symptoms, 5 = disabling symptoms)

CONTACTS AND LOCATIONS:
Overall Officials: Georgios D Koukoulis, MD, PhD, Principal Investigator — General Hospital of Larissa
Locations (1):
- General Hospital Of Larissa, Larissa, Greece

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] HerniaSurge Group. International guidelines for groin hernia management. Hernia. 2018 Feb;22(1):1-165. doi: 10.1007/s10029-017-1668-x. Epub 2018 Jan 12. PMID 29330835